CLINICAL TRIAL: NCT04859517
Title: A Phase 2/3 Randomized, Double-blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of ADG20 in the Prevention of COVID-19 (EVADE)
Brief Title: Evaluation of ADG20 for the Prevention of COVID-19
Acronym: EVADE
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: All primary efficacy data has been collected and analyzed. Based on the safety data gathered to date, it has been determined that continued participation by study subjects would not yield any additional beneficial safety information.
Sponsor: Invivyd, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ADG20-PREV-001
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-04

CONDITIONS: COVID-19
Keywords: Adintrevimab, ADG20, COVID-19, prevention, prophylaxis
MeSH Terms: conditions — COVID-19 | interventions — ADG20

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator, participant and sponsor personnel involved in study intervention and study evaluation will remain blinded to each participant's assigned study treatment throughout the course of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ADG20 (Experimental): Participants will be dosed on Day 1 with ADG20 IM
  Interventions: Drug: ADG20
- Placebo (Placebo Comparator): Participants will be dosed on Day 1 with placebo IM
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADG20 — Single dose of ADG20
  Arms: ADG20
Drug: Placebo — Single dose of placebo
  Arms: Placebo

SUMMARY:
This placebo-controlled study is intended to evaluate ADG20's safety and ability to prevent COVID-19 infection.

DETAILED DESCRIPTION:
Phase 2/3, multicenter, double-blind, placebo-controlled, randomized study of the mAb ADG20 in the prevention of symptomatic COVID-19 in adults and adolescents with no known history of SARS-CoV-2 infection but whose circumstances place them at increased risk of acquiring SARS-CoV-2 infection and developing symptomatic COVID-19. This objective was independently evaluated in a cohort of participants with reported recent exposure to an individual diagnosed with a SARS-CoV-2 infection (post-exposure prophylaxis) and in a cohort of participants with no reported exposure to SARS-CoV-2 (pre-exposure prophylaxis). These cohorts included participants whose advanced age (≥55 years old) or health status placed them at risk for severe COVID-19 or COVID-19 complications.

ELIGIBILITY:
Inclusion Criteria:

* Tests negative for current or previous SARS-CoV-2 infection by RT-PCR and serology (Pre-exposure population only)
* Is at high risk of SARS-CoV-2 infection as assessed by the Investigator:

  1. Post-exposure population: exposure to an individual with a diagnosis of SARS-CoV-2 infection (index case). Note: Participants with recent exposure to a laboratory-confirmed index case must be asymptomatic and randomized within 5 days (120 hours) of collection of the index case's positive SARS-CoV-2 diagnostic test.
  2. Pre-exposure population: Occupational, housing, recreational and/or social conditions that are likely to increase risk of exposure to SARS-CoV-2.
* Agrees to defer receipt of COVID-19 vaccination for minimum of 180 days (6 months) after dosing

Exclusion Criteria:

* Has received (1) a SARS-CoV-2 vaccine, (2) mAb or (3) convalescent plasma from a person who has recovered from COVID-19 or prior participation in SARS-CoV2 vaccine, convalescent plasma, or mAb clinical trial any time prior to participation in the study.
* Receipt of any investigational product within 30 days or 5 half lives before the day of enrollment.
* Is acutely ill or febrile 72 hours before or at Screening or has other COVID-19 symptoms including cough, fatigue, muscle or body aches, headache, or loss of taste or smell. Fever is defined as a body temperature ≥38.0°C (≥100.4°F).
* Has received or plans to receive a non-COVID-19 vaccine within 28 days before or after dosing (except for seasonal influenza vaccine, which is not permitted within 14 days before or after dosing).

NOTE: Other protocol defined inclusion/exclusion criteria apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2582 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (89):
- United States (63):
  - Invivyd Investigative Site, Birmingham, Alabama
  - Invivyd Investigative Site, Tucson, Arizona
  - Invivyd Investigative Site, Fayetteville, Arkansas
  - Invivyd Investigative Site, North Little Rock, Arkansas
  - Invivyd Investigative Site, Banning, California
  - Invivyd Investigative Site, Chula Vista, California
  - Invivyd Investigative Site, Culver City, California
  - Invivyd Investigative Site, Escondido, California
  - Invivyd Investigative Site, Fullerton, California
  - Invivyd Investigative Site, Long Beach, California
  - Invivyd Investigative Site, Los Angeles, California
  - Invivyd Investigative Site, Modesto, California
  - Invivyd Investigative Site, Palm Springs, California
  - Invivyd Investigative Site, San Diego, California
  - Invivyd Investigative Site, Clearwater, Florida
  - Invivyd Investigative Site, Edgewater, Florida
  - Invivyd Investigative Site, Hialeah, Florida
  - Invivyd Investigative Site, Miami, Florida
  - Invivyd Investigative Site, Mt. Dora, Florida
  - Invivyd Investigative Site, North Miami Beach, Florida
  - Invivyd Investigative Site, Ormond Beach, Florida
  - Invivyd Investigative Site, Pembroke Pines, Florida
  - Invivyd Investigative Site, Sunrise, Florida
  - Invivyd Investigative Site, Tampa, Florida
  - Invivyd Investigative Site, The Villages, Florida
  - Invivyd Investigative Site, West Palm Beach, Florida
  - Invivyd Investigative Site, Hinesville, Georgia
  - Invivyd Investigative Site, Lawrenceville, Georgia
  - Invivyd Investigative Site, Pearl City, Hawaii
  - Invivyd Investigative Site, Chicago, Illinois
  - Invivyd Investigative Site, Oak Brook, Illinois
  - Invivyd Investigative Site, Owensboro, Kentucky
  - Invivyd Investigative Site, Marrero, Louisiana
  - Invivyd Investigative Site, New Orleans, Louisiana
  - Invivyd Investigative Site, Rockville, Maryland
  - Invivyd Investigative Site, Burlington, Massachusetts
  - Invivyd Investigative Site, Caro, Michigan
  - Invivyd Investigative Site, Grosse Pointe Woods, Michigan
  - Invivyd Investigative Site, Missoula, Montana
  - Invivyd Investigative Site, Albuquerque, New Mexico
  - Invivyd Investigative Site, New York, New York
  - Invivyd Investigative Site, Charlotte, North Carolina
  - Invivyd Investigative Site, Shelby, North Carolina
  - Invivyd Investigative Site, Beachwood, Ohio
  - Invivyd Investigative Site, Cincinnati, Ohio
  - Invivyd Investigative Site, Dresden, Ohio
  - Invivyd Investigative Site, Middleburg Heights, Ohio
  - Invivyd Investigative Site, Yukon, Oklahoma
  - Invivyd Investigative Site, Medford, Oregon
  - Invivyd Investigative Site, West Columbia, South Carolina
  - Invivyd Investigative Site, Jackson, Tennessee
  - Invivyd Investigative Site, Milan, Tennessee
  - Invivyd Investigative Site, Nashville, Tennessee
  - Invivyd Investigative Site, Beaumont, Texas
  - Invivyd Investigative Site, College Station, Texas
  - Invivyd Investigative Site, Corpus Christi, Texas
  - Invivyd Investigative Site, Houston, Texas
  - Invivyd Investigative Site, Hurst, Texas
  - Invivyd Investigative Site, Mesquite, Texas
  - Invivyd Investigative Site, Sugar Land, Texas
  - Invivyd Investigative Site, St. George, Utah
  - Invivyd Investigative Site, West Jordan, Utah
  - Invivyd Investigative Site, Richmond, Virginia
- Argentina (6):
  - Invivyd Investigative Site, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Invivyd Investigative Site, Mar del Plata, Buenos Aires
  - Invivyd Investigative Site, Munro, Buenos Aires
  - Invivyd Investigative Site, Ramos Mejía, Buenos Aires
  - Invivyd Investigative Site, Rosario, Santa Fe Province
  - Invivyd Investigative Site, Rosario, Sante Fe
- Czechia (3):
  - Invivyd Investigative Site, Ostrava
  - Invivyd Investigative Site, Prague
  - Invivyd Investigative Site, Rychnov nad Kněžnou
- Georgia (4):
  - Invivyd Investigative Site, Batumi
  - Invivyd Investigative Site, Kutaisi
  - Invivyd Investigative Site, Rustavi
  - Invivyd Investigative Site, Tbilisi
- Invivyd Investigative Site, Berlin, Germany
- Invivyd Investigative Site, Chisinau, Moldova
- Poland (8):
  - Invivyd Investigative Site, Kajetany
  - Invivyd Investigative Site, Lodz
  - Invivyd Investigative Site, Lublin
  - Invivyd Investigative Site, Siedlce
  - Invivyd Investigative Site, Skierniewice
  - Invivyd Investigative Site, Swidnica
  - Invivyd Investigative Site, Warsaw
  - Invivyd Investigative Site, Zamość
- Invivyd Investigative Site, Bucharest, Romania
- Ukraine (2):
  - Adagio Investigative Site, Kyiv
  - Invivyd Investigative Site, Kyiv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ison MG, Weinstein DF, Dobryanska M, Holmes A, Phelan AM, Li Y, Gupta D, Narayan K, Tosh K, Hershberger E, Connolly LE, Yalcin I, Campanaro E, Hawn P, Schmidt P; EVADE Study Group. Prevention of COVID-19 Following a Single Intramuscular Administration of Adintrevimab: Results From a Phase 2/3 Randomized, Double-Blind, Placebo-Controlled Trial (EVADE). Open Forum Infect Dis. 2023 Jun 13;10(7):ofad314. doi: 10.1093/ofid/ofad314. eCollection 2023 Jul. PMID 37496612
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Groups:
- ADG20 IM - Cohort A: ADG20 IM - Cohort A is a post-exposure prophylaxis (PEP) arm where participants with no known history of SARS-CoV-2 infection and reported recent exposure (within 5 days) to SARS-CoV-2 were dosed with a single dose of ADG20 IM on Day 1.
- Placebo IM - Cohort A: Placebo IM - Cohort A is a post-exposure prophylaxis (PEP) arm where participants with no known history of SARS-CoV-2 infection and reported recent exposure (within 5 days) to SARS-CoV-2 were dosed with a single dose of placebo IM on Day 1.
- ADG20 IM - Cohort B: ADG20 IM - Cohort B is a pre-exposure prophylaxis (PrEP) arm where participants with no known history of SARS-CoV-2 infection and no known recent exposure to SARS-CoV-2 but whose circumstances put them at increased risk of exposure to SARS-CoV-2 were dosed with a single dose of ADG20 IM on Day 1.
- Placebo IM - Cohort B: Placebo IM - Cohort B is a pre-exposure prophylaxis (PrEP) arm where participants with no known history of SARS-CoV-2 infection and no known recent exposure to SARS-CoV-2 but whose circumstances put them at increased risk of exposure to SARS-CoV-2 were dosed with a single dose of placebo IM on Day 1.
Period: Overall Study
Arm/Group | ADG20 IM - Cohort A | Placebo IM - Cohort A | ADG20 IM - Cohort B | Placebo IM - Cohort B
Started | 245 | 242 | 1048 | 1047
Completed | 32 | 35 | 226 | 236
Not Completed | 213 | 207 | 822 | 811

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ADG20 IM - Cohort A | Placebo IM - Cohort A | ADG20 IM - Cohort B | Placebo IM - Cohort B | Total
Number analyzed (Participants) | 245 | 242 | 1048 | 1047 | 2582
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 2 | 7 | 2 | 16
  Between 18 and 65 years | 209 | 220 | 942 | 923 | 2294
  >=65 years | 31 | 20 | 99 | 122 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (15.61) | 45.4 (14.52) | 46.5 (13.90) | 47.1 (14.10) | 46.8 (14.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 120 | 508 | 522 | 1273
  Male | 122 | 122 | 540 | 525 | 1309
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 146 | 143 | 217 | 248 | 754
  Not Hispanic or Latino | 99 | 99 | 785 | 751 | 1734
  Unknown or Not Reported | 0 | 0 | 46 | 48 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 5 | 12 | 17
  Asian | 0 | 0 | 10 | 8 | 18
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 6 | 6 | 13
  Black or African American | 29 | 30 | 168 | 182 | 409
  White | 214 | 210 | 821 | 803 | 2048
  More than one race | 0 | 1 | 15 | 11 | 27
  Unknown or Not Reported | 1 | 1 | 23 | 25 | 50
Region of Enrollment [Number; unit: participants]
  Argentina | 0 | 1 | 6 | 7 | 14
  Romania | 43 | 36 | 0 | 0 | 79
  United States | 180 | 180 | 870 | 868 | 2098
  Czechia | 0 | 0 | 3 | 5 | 8
  Ukraine | 22 | 25 | 82 | 81 | 210
  Poland | 0 | 0 | 17 | 16 | 33
  Moldova | 0 | 0 | 5 | 2 | 7
  Georgia | 0 | 0 | 65 | 68 | 133

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With RT-PCR Confirmed Symptomatic COVID-19 (PEP)
Description: RT-PCR-confirmed symptomatic COVID-19 is determined by a positive central or local (in the absence of central test) RT-PCR test from a nasopharyngeal or saliva sample accompanied by protocol-defined COVID-19 symptoms occurring within 14 days from the sample collection date. Any COVID-19-related hospitalization with a positive local SARS-CoV-2 test (within 14 days) or all-cause death are counted toward the endpoint.
Time Frame: Day 1 through Day 28 or emergence of Omicron (15-Dec-2021), whichever is earlier
Population: Participants in the pre-Omicron modified Full Analysis Set-1 (mFAS-1): participants without current SARS-CoV-2 infection at baseline based on central tests (baseline RT-PCR-negative regardless of serostatus) randomized on or prior to 30-Nov-2021, allowing participants to be followed a minimum of 2 weeks through 15-Dec-2021 when Omicron became the predominant variant.
Measure: Count of Participants; unit: Participants
Groups:
- ADG20 IM - Cohort A: ADG20 IM - Cohort A is a post-exposure prophylaxis (PEP) arm where participants with no known history of SARS-CoV-2 infection and reported recent exposure (within 5 days) to SARS-CoV-2 were administered a single dose of ADG20 IM on Day 1.
- Placebo IM - Cohort A: Placebo IM - Cohort A is a post-exposure prophylaxis (PEP) arm where participants with no known history of SARS-CoV-2 infection and reported recent exposure (within 5 days) to SARS-CoV-2 were administered a single dose of placebo IM on Day 1.
Arm/Group | ADG20 IM - Cohort A | Placebo IM - Cohort A
Number analyzed (Participants) | 175 | 176
Participants | 3 | 12
Statistical Analysis 1: Comparison: ADG20 IM - Cohort A vs Placebo IM - Cohort A; Test type: Superiority; p = 0.0123, Regression, Logistic; Risk Difference (RD) = -5.0, 95% CI 2-sided [-8.87 to -1.08]; A statistical method described in Ge et al. (2011) was used to compute a population-level estimate for the treatment difference (in terms of difference in proportion) with adjustment for the pre-defined prognostic factors. The variance of the estimated treatment difference or relative risk reduction was estimated using the delta method

2. Primary Outcome: Percentage of Participants With RT-PCR Confirmed Symptomatic COVID-19 (PrEP)
Description: as for outcome 1
Time Frame: Day 1 through 3 Months or emergence of Omicron (15-Dec-2021), whichever is earlier
Population: Participants in the pre-Omicron modified Full Analysis Set (mFAS): participants without prior or current SARS-CoV-2 infection at baseline based on central tests (baseline RT-PCR-negative and seronegative) randomized on or prior to 30-Nov-2021, allowing participants to be followed a minimum of 2 weeks through 15-Dec-2021 when Omicron became the predominant variant.
Measure: Count of Participants; unit: Participants
Groups:
- ADG20 IM - Cohort B: ADG20 IM - Cohort B is a pre-exposure prophylaxis (PrEP) arm where participants with no known history of SARS-CoV-2 infection and no known recent exposure to SARS-CoV-2 but whose circumstances put them at increased risk of exposure to SARS-CoV-2 were administered a single dose of ADG20 IM on Day 1.
- Placebo IM - Cohort B: Placebo IM - Cohort B is a pre-exposure prophylaxis (PrEP) arm where participants with no known history of SARS-CoV-2 infection and no known recent exposure to SARS-CoV-2 but whose circumstances put them at increased risk of exposure to SARS-CoV-2 were administered a single dose of placebo IM on Day 1.
Arm/Group | ADG20 IM - Cohort B | Placebo IM - Cohort B
Number analyzed (Participants) | 752 | 728
Participants | 12 | 40
Statistical Analysis 1: Comparison: ADG20 IM - Cohort B vs Placebo IM - Cohort B; Test type: Superiority; p < 0.0001, Regression, Logistic; Risk Difference (RD) = -3.9, 95% CI 2-sided [-5.75 to -2.01]

3. Primary Outcome: Solicited Injection Site Reactions (PEP, PrEP)
Description: Percentage of participants with at least one solicited injection site reaction
Time Frame: Day 1 through Day 4
Population: Participants who received any amount of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM - Cohort A | Placebo IM - Cohort A | ADG20 IM - Cohort B | Placebo IM - Cohort B
Number analyzed (Participants) | 240 | 241 | 1001 | 1001
Participants | 12 | 7 | 75 | 73

4. Primary Outcome: Participants With at Least 1 Treatment Emergent Adverse Events (PEP, PrEP)
Description: Any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment; includes solicited injection site reactions
Time Frame: Day 1 through 14 Months or 25Jul2022, whichever is earlier
Population: Participants who received any amount of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM - Cohort A | Placebo IM - Cohort A | ADG20 IM - Cohort B | Placebo IM - Cohort B
Number analyzed (Participants) | 240 | 241 | 1001 | 1001
Participants | 42 | 51 | 399 | 362

5. Secondary Outcome: Percentage of Participants With RT-PCR Confirmed Symptomatic COVID-19 (PEP)
Description: RT-PCR-confirmed symptomatic COVID-19 is determined by a positive central or local (in the absence of central test) RT-PCRtest from a nasopharyngeal or saliva sample accompanied by protocol-defined COVID-19 symptoms occurring within 14 days from the sample collection date. Any COVID-19-related hospitalization with a positive local SARS-CoV-2 test (within 14 days) or all-cause death are counted toward the endpoint.
Time Frame: Day 1 through Day 28 or emergence of Omicron (15-Dec-2021), whichever is earlier
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM - Cohort A | Placebo IM - Cohort A
Number analyzed (Participants) | 76 | 79
Participants | 1 | 7
Statistical Analysis 1: Comparison: ADG20 IM - Cohort A vs Placebo IM - Cohort A; Test type: Superiority; p = 0.0153, Regression, Logistic; Standardized Risk Difference = -7.6, 95% CI 2-sided [-13.74 to -1.46]; [other analysis details as in outcome 1, analysis 1]

6. Secondary Outcome: Percentage of Participants With SARS-CoV-2 Infection (Asymptomatic or Symptomatic) as Determined by Positive RT-PCR or Serology (PEP)
Description: Participants with RT-PCR-confirmed symptomatic COVID-19 (protocol defined COVID-19 symptoms occurring within 14 days from the sample collection date of a positive central or local [in the absence of central test] RT-PCR, any COVID-19-related hospitalization with a positive local SARS-CoV-2 test [within 14 days], or all-cause death), central RT-PCR-confirmed SARS-CoV-2 infection, or central serology-confirmed SARS-CoV-2 infection with negative central serology at baseline.
Time Frame: Day 1 through Day 28 or emergence of Omicron (15-Dec-2021), whichever is earlier
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM - Cohort A | Placebo IM - Cohort A
Number analyzed (Participants) | 175 | 176
Participants | 6 | 14
Statistical Analysis 1: Comparison: ADG20 IM - Cohort A vs Placebo IM - Cohort A; Test type: Superiority; p = 0.0612, Regression, Logistic; Risk Difference (RD) = -4.4, 95% CI 2-sided [-9.03 to 0.21]; [other analysis details as in outcome 1, analysis 1]

7. Secondary Outcome: Percentage of Participants With Asymptomatic SARS-CoV-2 Infection as Determined by RT-PCR (PEP)
Description: Defined as having a central RT-qPCR-confirmed SARS-CoV-2 infection without having an RT-PCR-confirmed symptomatic COVID-19 outcome
Time Frame: Day 1 through Day 28 or emergence of Omicron (15-Dec-2021), whichever is earlier
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM - Cohort A | Placebo IM - Cohort A
Number analyzed (Participants) | 175 | 176
Participants | 3 | 1

8. Secondary Outcome: Percentage of Participants With Asymptomatic SARS-CoV-2 Infection as Determined by Serology (PEP)
Description: Defined as having a central serology-confirmed SARS-CoV-2 infection (with a negative central serology test sample at baseline) and without having an RT-PCR-confirmed symptomatic COVID-19 outcome (including COVID-19-related hospitalization and all-cause death)
Time Frame: Day 1 through Day 28 or emergence of Omicron (15-Dec-2021), whichever is earlier
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM - Cohort A | Placebo IM - Cohort A
Number analyzed (Participants) | 175 | 176
Participants | 0 | 1

9. Secondary Outcome: Percentage of Participants With Asymptomatic SARS-CoV-2 Infection as Determined by Serology (PrEP)
Description: as for outcome 8
Time Frame: Day 1 through 6 Months or emergence of Omicron (15-Dec-2021), whichever is earlier
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM - Cohort B | Placebo IM - Cohort B
Number analyzed (Participants) | 752 | 728
Participants | 10 | 18

10. Secondary Outcome: SARS-CoV-2 Viral Load as Assessed by RT-qPCR Change From Baseline in Asymptomatic Participants (PEP)
Description: Asymptomatic SARS-CoV-2 infection confirmed by RT-qPCR from nasal swab collected at Day 8 and Day 15. Viral load values reported as detected but below the lower quantification of the PCR assay (< 714 copies/mL) are imputed with half the lower limit of quantification of the PCR assay (i.e., 357 copies/mL = 2.55 log10 copies/mL). Viral load values reported as > 7.1×10^7 copies/mL are imputed with 7.1×10^7 copies/mL (i.e., 7.85 log10 copies/mL).
Time Frame: Day 1 through Day 28 or emergence of Omicron (15-Dec-2021), whichever is earlier
Population: Participants with RT-qPCR-confirmed asymptomatic SARS-CoV-2 infection in the pre-Omicron modified Full Analysis Set-1 (mFAS-1): participants without current SARS-CoV-2 infection at baseline based on central tests (baseline RT-PCR-negative regardless of serostatus) randomized on or prior to 30-Nov-2021, allowing participants to be followed a minimum of 2 weeks through 15-Dec-2021 when Omicron became the predominant variant.
Measure: Mean (Standard Deviation); unit: Viral load (log10 copies/mL)
Arm/Group | ADG20 IM - Cohort A | Placebo IM - Cohort A
Number analyzed (Participants) | 3 | 1
Viral load (log10 copies/mL)
  Day 8 | 2.96 (4.186) | 0 (0)
  Day 15 | 2.15 (1.985) | 3.16

11. Secondary Outcome: Percentage of Participants With RT-PCR Confirmed Mild, Moderate, or Severe/Critical COVID-19 (PEP)
Description: Maximum severity assessed from COVID-19-like illness (CLI) Day 1 through CLI Day 28. COVID-19-related hospitalizations or COVID-19-related deaths from CLI Day 1 to CLI Day 28 are categorized as severe/critical.
Time Frame: Day 1 through Day 28 or emergence of Omicron (15-Dec-2021), whichever is earlier
Population: Participants with RT-PCR confirmed symptomatic COVID-19 in the pre-Omicron modified Full Analysis Set-1 (mFAS-1): participants without current SARS-CoV-2 infection at baseline based on central tests (baseline RT-PCR-negative regardless of serostatus) randomized on or prior to 30-Nov-2021, allowing participants to be followed a minimum of 2 weeks through 15-Dec-2021 when Omicron became the predominant variant.
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM - Cohort A | Placebo IM - Cohort A
Number analyzed (Participants) | 3 | 12
Participants
  Cohort A (PEP) Mild | 3 | 7
  Cohort A (PEP) Moderate | 0 | 2
  Cohort A (PEP) Severe/Critical | 0 | 3

12. Secondary Outcome: Percentage of Participants With RT-PCR Confirmed Mild, Moderate, or Severe/Critical COVID-19 (PrEP)
Description: as for outcome 11
Time Frame: Day 1 through 3 Months or emergence of Omicron (15-Dec-2021), whichever is earlier
Population: Participants with RT-PCR confirmed symptomatic COVID-19 in the pre-Omicron modified Full Analysis Set (mFAS): participants without prior or current SARS-CoV-2 infection at baseline based on central tests (baseline RT-PCR-negative and seronegative) randomized on or prior to 30-Nov-2021, allowing participants to be followed a minimum of 2 weeks through 15-Dec-2021 when Omicron became the predominant variant.
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM - Cohort B | Placebo IM - Cohort B
Number analyzed (Participants) | 12 | 40
Participants
  Cohort B (PrEP) Mild | 7 | 14
  Cohort B (PrEP) Moderate | 4 | 19
  Cohort B (PrEP) Severe/Critical | 1 | 7

13. Secondary Outcome: Percentage of Participants With at Least 1 COVID-19 Related Medically Attended Outpatient Visit (PEP)
Description: Physician office, telemedicine, emergency room or urgent care center visits in participants with RT-PCR-confirmed symptomatic COVID-19 events, defined as having a central RT-PCR-confirmed SARS-CoV-2 infection with COVID-19 symptoms occurring within 14 days from the positive RT-PCR test sample collection, COVID-19-related hospitalization with a positive local or central SARS-CoV-2 test within 14 days, or all-cause death.
Time Frame: Day 1 through Day 28 or emergence of Omicron (15-Dec-2021), whichever is earlier
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM - Cohort A | Placebo IM - Cohort A
Number analyzed (Participants) | 3 | 12
Participants | 0 | 3

14. Secondary Outcome: Percentage of Participants With at Least 1 COVID-19 Related Medically Attended Outpatient Visit (PrEP)
Description: Physician office, telemedicine, emergency room or urgent care center visits in participants with RT-PCR confirmed symptomatic COVID-19, defined as having a central RT-PCR-confirmed SARS-CoV-2 infection with COVID-19 symptoms occurring within 14 days from the positive RT-PCR test sample collection, COVID-19-related hospitalization with a positive local or central SARS-CoV-2 test within 14 days, or all-cause death.
Time Frame: Day 1 through 3 Months or emergence of Omicron (15-Dec-2021), whichever is earlier
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM - Cohort B | Placebo IM - Cohort B
Number analyzed (Participants) | 12 | 40
Participants | 1 | 6

15. Secondary Outcome: Percentage of Participants With a COVID-19 Related Hospitalization (PEP)
Time Frame: Through 28 Days from COVID-19-like illness initial visit (CLI Day 1)
Population: Participants with RT-PCR confirmed symptomatic COVID-19 through Day 28 in the pre-Omicron modified Full Analysis Set-1 (mFAS-1): participants without current SARS-CoV-2 infection at baseline based on central tests (baseline RT-PCR-negative regardless of serostatus) randomized on or prior to 30-Nov-2021, allowing participants to be followed a minimum of 2 weeks through 15-Dec-2021 when Omicron became the predominant variant.
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM - Cohort A | Placebo IM - Cohort A
Number analyzed (Participants) | 3 | 12
Participants | 0 | 3

16. Secondary Outcome: Percentage of Participants With a COVID-19 Related Hospitalization (PrEP)
Time Frame: Through 28 days from COVID-19-like illness initial visit (CLI Day 1)
Population: Participants with RT-PCR confirmed symptomatic COVID-19 through Month 3 in the pre-Omicron modified Full Analysis Set (mFAS): participants without prior or current SARS-CoV-2 infection at baseline based on central tests (baseline RT-PCR-negative and seronegative) randomized on or prior to 30-Nov-2021, allowing participants to be followed a minimum of 2 weeks through 15-Dec-2021 when Omicron became the predominant variant.
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM - Cohort B | Placebo IM - Cohort B
Number analyzed (Participants) | 12 | 40
Participants | 1 | 6

17. Secondary Outcome: COVID-19 Related Mortality (PEP)
Time Frame: Through 28 Days from COVID-19-like illness initial visit (CLI Day 1)
Population: Participants with RT- PCR confirmed symptomatic COVID-19 in the pre-Omicron modified Full Analysis Set-1 (mFAS-1): participants without current SARS-CoV-2 infection at baseline based on central tests (baseline RT-PCR-negative regardless of serostatus) randomized on or prior to 30-Nov-2021, allowing participants to be followed a minimum of 2 weeks through 15-Dec-2021 when Omicron became the predominant variant.
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM - Cohort A | Placebo IM - Cohort A
Number analyzed (Participants) | 3 | 12
Participants | 0 | 0

18. Secondary Outcome: COVID-19 Related Mortality (PrEP)
Time Frame: Through 28 Days from COVID-19-like illness initial visit (CLI Day 1)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM - Cohort B | Placebo IM - Cohort B
Number analyzed (Participants) | 12 | 40
Participants | 0 | 1

19. Secondary Outcome: All-Cause Mortality (PEP)
Time Frame: Through 28 Days from COVID-19-like illness initial visit (CLI Day 1)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM - Cohort A | Placebo IM - Cohort A
Number analyzed (Participants) | 3 | 12
Participants | 0 | 0

20. Secondary Outcome: All-Cause Mortality (PrEP)
Time Frame: Through 28 Days from COVID-19-like illness initial visit (CLI Day 1)
Population: Participants with RT-PCR confirmed symptomatic COVID-19 through Month 3 in the pre-Omicron modified Full Analysis Set (mFAS): PrEP participants without prior or current SARS-CoV-2 infection at baseline based on central tests (baseline RT-PCR-negative and seronegative) randomized on or prior to 30-Nov-2021, allowing participants to be followed a minimum of 2 weeks through 15-Dec-2021 when Omicron became the predominant variant.
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM - Cohort B | Placebo IM - Cohort B
Number analyzed (Participants) | 12 | 40
Participants | 0 | 1

21. Secondary Outcome: Viral Load as Assessed by RT-qPCR in Participants With Confirmed Symptomatic COVID-19 (PEP)
Description: Viral load from COVID-19-like illness (CLI) Day 1 sample. Viral load values reported as detected but below the lower quantification of the PCR assay (< 714 copies/mL) are imputed with half the lower limit of quantification of the PCR assay (i.e., 357 copies/mL = 2.55 log10 copies/mL). Viral load values reported as > 7.1×10^7 copies/mL are imputed with 7.1×10^7 copies/mL (i.e., 7.85 log10 copies/mL).
Time Frame: Positive CLI Day 1 sample through Day 28 or emergence of Omicron (15-Dec-2021), whichever is earlier
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | ADG20 IM - Cohort A | Placebo IM - Cohort A
Number analyzed (Participants) | 3 | 12
log10 copies/mL | 2.43 (2.372) | 5.74 (2.689)

22. Secondary Outcome: Viral Load as Assessed by RT-qPCR in Participants With Confirmed Symptomatic COVID-19 (PrEP)
Description: as for outcome 21
Time Frame: Positive CLI Day 1 sample through 3 Months or emergence of Omicron (15-Dec-2021), whichever is earlier
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | ADG20 IM - Cohort B | Placebo IM - Cohort B
Number analyzed (Participants) | 12 | 40
Log10 copies/mL | 4.58 (2.730) | 6.58 (1.825)

23. Secondary Outcome: Assessment of PK Parameter: ADG20 Plasma Concentrations (PEP)
Description: PK samples collected at protocol-defined timepoints
Time Frame: Day 1 through 12 Months or end of study (11-Jan-2022), whichever is earlier
Population: Participants who received study drug and have measurable ADG20 concentration data for at least 2 post-injection time points
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | ADG20 IM - Cohort A
Number analyzed (Participants) | 52
ug/mL
  Day 8 | 36.3 (15.4)
  Day 28 | 33.6 (12.6)

24. Secondary Outcome: Assessment of PK Parameter: ADG20 Plasma Concentrations (PrEP)
Description: PK samples collected at protocol-defined timepoints
Time Frame: Day 1 through 12 Months or end of study (11-Jan-2022), whichever is earlier
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | ADG20 IM - Cohort B
Number analyzed (Participants) | 353
ug/mL
  Day 8 | 38.2 (14.7)
  Day 28 | 33.6 (12.5)

25. Secondary Outcome: Time From Randomization to First RT-PCR-confirmed Symptomatic COVID-19 (PEP)
Description: Outcome measure is presented as cumulative probability expressed in percentage. RT-PCR-confirmed symptomatic COVID-19 event is defined as having a central RT-PCR-confirmed SARS-CoV-2 infection with COVID-19 symptoms occurring within 14 days from the positive RT-PCR test sample collection, COVID-19-related hospitalization with a positive local or central SARS-CoV-2 test within 14 days, or all-cause death.
Time Frame: An average of 2 months up to 7 months through cutoff date prior to emergence of Omicron (15-Dec-2021)
Population: as for outcome 1
Measure: Number; unit: Percent probability
Arm/Group | ADG20 IM - Cohort A | Placebo IM - Cohort A
Number analyzed (Participants) | 175 | 176
Percent probability
  Day 28 | 1.74 | 7.01
  Day 60 | 1.74 | 7.84
  Day 90 | 1.74 | 7.84
Statistical Analysis 1: Comparison: ADG20 IM - Cohort A vs Placebo IM - Cohort A; Test type: Superiority; p = 0.0077, Log Rank; Hazard Ratio (HR) = 0.22, 95% CI 2-sided [0.06 to 0.76]

26. Secondary Outcome: Time From Randomization to First RT-PCR-confirmed Symptomatic COVID-19 (PrEP)
Description: as for outcome 25
Time Frame: An average of 2.5 months up to 7.5 months through cutoff date prior to emergence of Omicron (15-Dec-2021)
Population: as for outcome 2
Measure: Number; unit: Percent probability
Arm/Group | ADG20 IM - Cohort B | Placebo IM - Cohort B
Number analyzed (Participants) | 752 | 728
Percent probability
  Day 28 | 0.96 | 2.32
  Day 60 | 1.31 | 5.64
  Day 90 | 2.01 | 7.26
Statistical Analysis 1: Comparison: ADG20 IM - Cohort B vs Placebo IM - Cohort B; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.27, 95% CI 2-sided [0.14 to 0.49]

ADVERSE EVENTS:
Time Frame: Baseline through Month 14 or end of study (11-Jan-2022), whichever is earlier
Description: Safety analysis set: All participants who received any amount of study drug
Arm/Group | ADG20 IM - Cohort A | Placebo IM - Cohort A | ADG20 IM - Cohort B | Placebo IM - Cohort B
All-Cause Mortality (participants affected / at risk) | 0/240 | 2/241 | 3/1001 | 6/1001
Serious Adverse Events (participants affected / at risk) | 4/240 | 8/241 | 46/1001 | 46/1001
Other Adverse Events (participants affected / at risk) | 0/240 | 0/241 | 126/1001 | 123/1001
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADG20 IM - Cohort A (N=240) | Placebo IM - Cohort A (N=241) | ADG20 IM - Cohort B (N=1001) | Placebo IM - Cohort B (N=1001)
COVID-19 pneumonia (Infections and infestations) | 1 | 4 | 1 | 9
Pneumonia (Infections and infestations) | 1 | 0 | 4 | 2
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 3 | 6 — COVID-19 only captured as an AE if serious criteria met
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Testicular abscess (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 1
Hepatitis A (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis orbital (Infections and infestations) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Shrapnel wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Musculoskeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Meniscus cyst (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Non-small cell lung cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 2 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0
Substance-induced mood disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Schizoaffective disorder depressive type (Psychiatric disorders) | 0 | 0 | 0 | 1
Schizoaffective disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Delirium tremens (Psychiatric disorders) | 0 | 0 | 1 | 0
Small intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Myelopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1
Visual field defect (Eye disorders) | 0 | 0 | 0 | 1
Angle closure glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ADG20 IM - Cohort A (N=240) | Placebo IM - Cohort A (N=241) | ADG20 IM - Cohort B (N=1001) | Placebo IM - Cohort B (N=1001)
Injection site pain (General disorders) | NA | NA | 76 | 84
Influenza like illness (General disorders) | NA | NA | 59 | 46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT04859517/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/17/NCT04859517/SAP_001.pdf